CLINICAL TRIAL: NCT04772651
Title: Mediterranean Diet and the Microbiota Gut Brain Axis- Does Diet Interact With the Function of Vagal Nerve in Major Depression?
Brief Title: Mediterranean Diet and the Microbiota Gut Brain Axis in Major Depression
Acronym: MeDiVa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EK 1087 ex 2021
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Depression
Keywords: nutrition; mediterranean diet; vagal function; heart rate variability
MeSH Terms: conditions — Depression | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet and dietary coaching (Experimental): Patients receive 3 Mediterranean meals a day for 4 weeks and dietary coaching sessions (á 50 minutes once a week for 4 weeks)
  Interventions: Other: Mediterranean Diet; Other: dietary coaching
- Diet as usual and psychoeducation for depression (Placebo Comparator): Patients receive normal hospital diet with 3 meals a day for 4 weeks and psychoeducation sessions (á 50 minutes once a week for 4 weeks)
  Interventions: Other: Normal hospital diet; Other: Psychoeducation on depression

INTERVENTIONS:
Other: Mediterranean Diet — Diet meeting the requirements for mediterranean style (rich in vegetables, fruit, olive oil, fish) (Davis et al., 2015)
  Arms: Mediterranean Diet and dietary coaching
Other: Normal hospital diet — Normal hospital diet
  Arms: Diet as usual and psychoeducation for depression
Other: dietary coaching — dietary coaching
  Arms: Mediterranean Diet and dietary coaching
Other: Psychoeducation on depression — Psychoeducation on depression (50minutes once a week for 4 weeks)
  Arms: Diet as usual and psychoeducation for depression

SUMMARY:
The purpose of this study is to assess the efficacy of a Mediterranean diet on the function of the vagal nerve in patients with depression.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be screened for eligibility. Subjects meeting the inclusion criteria will be randomized in a group recieiving a Mediterranean diet (3 mediterranean meals a day) and dietary coaching (1 session per week for 4 weeks) or a group with conventional hospital food and psychoeducation on depression (1 session per week for 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* legally competent persons aged 18-80 years
* diagnosis of depression according to ICD-10 or DSM.

Exclusion Criteria:

* other neurologic or psychiatric disorders (epilepsy, brain tumor, head injury, head surgery, trauma)
* drug or alcohol dependency
* acute suicidality
* heart disorders, disorders of the circulatory system
* pregnancy and period of breastfeeding
* severe mental disability, dementia (MMST<20)
* autoimmune disorder, severe immunosuppression (Lupus, HIV, multiple sclerosis)
* therapy with antibiotics in the last month
* chronic laxative abuse
* acute infectious diarrhea
* GI surgeries (except appendectomy)
* regular intake of probiotics, antibiotics and food supplements (1 month before and during the study)
* food allergies or other food intolerances which are incompatible with a mediterranean diet
* vegetarians, vegans

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Vagal function | at study entry, after 7 days, after 4 weeks and after 3 months
  Vagal function measured by 24-hr ECG (logRSA, SDNN)

SECONDARY OUTCOMES:
Change of C-reactive protein (CRP) | at study entry, after 7 days, after 4 weeks and after 3 months
  CRP will be measured from serum samples at the Institute of laboratory diagnostics (Cobas analyzer)
Change in Interleukine-6 | at study entry, after 7 days, after 4 weeks and after 3 months
  Interleukine-6 will be measured from serum samples at the Institute of laboratory diagnostics
Change in Oxytocin | at study entry, after 7 days, after 4 weeks and after 3 months
  measured from serum samples with ELISA
Change of Gut microbiome | at study entry, after 7 days, after 4 weeks and after 3 months
  16S sequencing of a stool sample, gut microbiome data will be analyzed with QIIME2 with regard to diversity metrices (alpha-diversity, beta-diversity) and differential bacterial abundance.
Change of Body mass Index | at study entry, after 7 days, after 4 weeks and after 3 months
  Weight will be measured with a calibrated scale, height will be measured with a non-expandable measuring tape. BMI will be calculated according to the formula [kg/m2].
Change in Hamilton Scale for Depression (HAMD) | at study entry, after 7 days, after 4 weeks and after 3 months
  Scale to rate severity of depressive symptoms; Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression
Change in Beck Depression Inventory (BDI) | at study entry, after 7 days, after 4 weeks and after 3 months
  Self-rated scale to rate severity of depressive symptoms; Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
Change in Pittsburgh Sleep Quality Inventory (PSQI) | at study entry, after 7 days, after 4 weeks and after 3 months
  Questionnaire to assess sleep quality; global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Change in Adult Attachment Scale | at study entry, after 7 days, after 4 weeks and after 3 months
  Questionnaire to assess attachment style in adults; The scale consists of 18 items scored on a 5 point likert-type scale. It measures adult attachment styles named "Secure", "Anxious" and "Avoidant", defined as:
  * Secure = high scores on Close and Depend subscales, low score on Anxiety subscale
  * Anxious = high score on Anxiety subscale, moderate scores on Close and Depend subscales
  * Avoidant = low scores on Close, Depend, and Anxiety subscales
Change in Wiener Ernährungsprotokoll | at study entry, after 7 days, after 4 weeks and after 3 months
  24-hr food recall
Change in Mediterranean Diet Score | at study entry, after 7 days, after 4 weeks and after 3 months
  Questionnaire rating the diet according to Mediterranean dietary style; three categories of adherence to the Mediterranean diet can be calculated (≤5, 6-9 and ≥10 points of the 14-item questionnaire)
Change in International Physical Acitivity Questionnaire | at study entry, after 7 days, after 4 weeks and after 3 months
  Questionnaire to rate physical activity; Physical activity is given in MET-minutes (METs are multiples of the resting metabolic rate)

IPD SHARING:
Plan to Share IPD: No